CLINICAL TRIAL: NCT06853041
Title: Etude randomisée contrôlée en Double-aveugle ESKAPE : ESKétamine Low-dose Versus kétamine Low-dose Pour la Douleur Aiguë sévère Aux Urgences, Comparaison Des Effets PsychodyslEptiques
Brief Title: ESKetamine Low-dose vs Ketamine Low-dose for Severe Acute Pain in Emergency Units, Comparison of PsychodyslEptic Effects
Acronym: ESKAPE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-PP-09
Record Dates: First submitted 2025-02-06; First posted 2025-02-28 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Esketamine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose esketamine (Experimental)
  Interventions: Drug: Esketamine
- low-dose ketamine (Active Comparator)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Esketamine — A single slow intravenous injection of low-dose esketamine (0.15 mg/kg) over 10 minutes using an infusion pump.
  Arms: low-dose esketamine
Drug: Ketamine — A single slow intravenous injection of low-dose ketamine (0,3 mg/kg) with an infusion pump, during 10 minutes
  Arms: low-dose ketamine

SUMMARY:
Almost 30% of painful patients in emergency departments (ED) describe their pain as severe (i.e. a Verbal Numerical Rating Score VNRS ≥ 6 on a scale ranging from 0 to 10). The management of such severe pain needs to be rapid and safe, and for this purpose intravenous (IV) morphine titration is still the gold-standard. However, morphine titration takes up considerable caregiver time, as patients need to be monitored and treated progressively with small quantities of morphine every 5 minutes until analgesia. This is sometimes difficult to reconcile with a saturating flow of patients, and overcrowding in ED is proven to significantly delay time-to-analgesia, and even lead to deleterious under-treatment. Finally, the opioid crisis is a major concern, explaining why strategies are being advocated to develop other ways of managing severe acute pain in the ED and to limit the use of opioids.

Recent studies show that ketamine administered in small IV doses ("low-dose" ketamine LDK: 0.2 to 0.3 mg/kg) possesses potent analgesic activity as well as interesting anti-hyperalgesic and anti-allodynic properties. Compared with morphine, LDK does not induce respiratory depression, but can sometimes induce disturbing psychodysleptic effects. These may include a sensation of unreality, fatigue, anxiety, dizziness or hallucinations. According to studies, 30-80% of LDK-treated patients experience psychodysleptic effects. However, two recent studies suggest that slow IV injections of LDK (over 10 minutes) may improve patient tolerance, although these slow infusions do not totally reduce this discomfort.

Pharmacologically, ketamine is a racemic mixture of 2 isomers: esketamine S(+), which is dextrorotatory, and arketamine R(-), which is levorotatory. In recent years, a new formulation containing only esketamine has been made available to hospitals in some northern European countries, and more recently in France. Esketamine appears to have twice the analgesic efficacy of racemic ketamine, and studies on healthy volunteers or in peri-operative settings suggest that it is also better tolerated psychologically than ketamine. For the moment, however, scientific data are lacking, and no comparative trial has yet been conducted in the ED setting. The investigators plan to conduct in their ED a prospective, single-center, randomized, double-blind study aiming to compare the tolerance and efficacy of esketamine versus racemic LDK in patients presenting with severe acute pain (VNRS ≥ 6/10).

DETAILED DESCRIPTION:
More than two-thirds of patients visiting emergency departments (ED) complain of acute pain, and of these, almost 30% describe their pain as severe (i.e. a Verbal Numerical Rating Score VNRS ≥ 6 on a scale ranging from 0 to 10). The management of such severe pain needs to be rapid, safe and adapted to the suspected underlying causative pathology. To achieve this, recommendations call for widespread use of intravenous (IV) morphine titration, which combines high analgesic efficacy with a good clinical safety profile (low risk of respiratory depression). However, the need to monitor patients and inject small quantities of morphine every 5 minutes until the patient is relieved takes up a considerable amount of caregiver time, which is sometimes difficult to reconcile with a saturating flow of patients. This growing problem of overcrowding in ED can lead to significant under-treatment and delays in analgesia. At the same time, the opioid crisis in the USA is beginning to affect other countries, which explains why certain strategies are being advocated to limit the use of opioids, and why researchers are attempting to develop other ways of managing severe acute pain in the ED. Recent studies show that ketamine administered in small IV doses ("low-dose" ketamine KLD: 0.2 to 0.3 mg/kg) possesses potent analgesic activity comparable to that of IV morphine. These analgesic qualities have been known for decades, and ketamine's unique non-competitive antagonism of the NMDA (N-methyl-D-aspartic) receptor also results in interesting anti-hyperalgesic and anti-allodynic properties. Compared with morphine, KLD does not induce the risk of respiratory depression, but can induce psychodysleptic effects that can sometimes be troublesome. These may include a sensation of unreality, fatigue, anxiety, dizziness or hallucinations. According to studies, 30 to 80% of patients treated with KLD experience a psychodysleptic effect. However, two recent studies suggest that slow IV injections of KLD (>10 min) may improve patient tolerance, although this slow injection may not significantly reduce this discomfort. Pharmacologically, ketamine is a racemic mixture of 2 isomers: esketamine S(+), which is dextrorotatory, and arketamine R(-), which is laevorotatory. In recent years, a new formulation containing only esketamine has been made available to hospitals in some northern European countries, and more recently in France. Esketamine appears to have twice the analgesic efficacy of racemic ketamine, and studies on healthy volunteers or in peri-operative settings suggest that it is also better tolerated psychologically than ketamine. For the moment, however, scientific data are lacking, and to our knowledge no comparative trial has yet been conducted in the ED setting. The prospective, single-center, randomized, double-blind study the investigators plan to conduct in the ED will compare the tolerance and efficacy of esketamine versus racemic LDK in patients presenting with severe acute pain (VNRS ≥ 6/10).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 or over,
* consulting our emergency department for a medical or traumatic pathology responsible for acute (less than 7 days old) and severe pain (greater than or equal to 6 on the Verbal Numerical Rating Scale, which has 11 levels from 0 = no pain to 10 = maximum imaginable pain).
* Free and informed consent given before the start of the trial.
* Patients affiliated to social security system.

Exclusion Criteria:

* Inability to quantify pain score ;
* proven or suspected intoxication (drug or alcohol) leading to consciousness disorders (Glasgow score less than or equal to 15) ;
* person under legal protection or deprived of liberty ;
* pregnant or breast-feeding patients ;
* known allergy to ketamine or esketamine ;
* history of drug addiction or dependence ;
* insufficiently controlled hyperthyroidism ;
* history of cerebral of myocardial infarction ;
* known severe heart failure ;
* existence of intracranial hypertension, glaucoma or ocular trauma ;
* unstable vital signs (systolic blood pressure < 90 mmHg or > 180, heart rate < 50 per minute or > 150, respiratory rate < 10 per minute or > 30) ;
* chronic treatment with aminophylline, theophylline or methylergometrine ;
* administration of morphine or another opioid within one hour of inclusion ;
* ongoing simultaneous participation in another study that could interfere with the treatment studied or the results of statistical analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing at least one psychodysleptic effect of the SERSDA (Side Effects Rating Scale for Dissociate Anesthetics) scale. | The time of initiation of the ketamine or esketamine infusion defines the minute 0 time point of the study. The presence of any of these 9 SERSDA items will be assessed by patients every 5 minutes from minute 0 to minute 0 + 60 minutes.
  The primary endpoint will be the proportion of patients experiencing at least one psychodysleptic effect, in the control group (ketamine IV 0.3 mg/kg) and in the active group (esketamine IV 0.15 mg/kg). Using the SERSDA (Side Effects Rating Scale for Dissociate Anesthetics) scale, the most widely used in studies, which comprises 9 items: fatigue, headache, dizziness, feeling of unreality, generalized feeling of discomfort, hearing changes, vision changes, mood change, hallucination.

SECONDARY OUTCOMES:
Intensity of the psychodysleptic effects described by patients. | The time of initiation of the ketamine or esketamine infusion defines the minute 0 time point of the study. The intensity of the psychodysleptic effects will be assessed by patients every 5 minutes from minute 0 to minute 0 + 60 minutes.
  For this secondary outcome, the 4 intensity items of the SERSDA (Side Effects Rating Scale for Dissociative Anesthetics) will be used : 1 = weak effect, 2 = moderate effect, 3 = troublesome effect and 4 = very troublesome effect.
Analgesic efficacy of the 2 molecules (ketamine or esketamine) | The time of initiation of the ketamine or esketamine infusion defines the minute 0 time point of the study. The intensity of the psychodysleptic effects will be assessed by patients every 5 minutes from minute 0 to minute 0 + 60 minutes.
  1. evolution of the Verbal Numercial Rating Score VNRS (scale from 0 "no pain" to 10 = "worst pain imainalbe") as a function of time 2. proportion of patients reporting pain relief (Verbal Numerical Rating Score VNRS ≤ 3/10) 3. proportion of patients needing additional analgesia ("rescue analgesia") which will be at the discretion of the physicians
Any other hemodynamic and respiratory adverse event | The time of initiation of the ketamine or esketamine infusion defines the minute 0 time point of the study. The intensity of the psychodysleptic effects will be assessed by patients every 5 minutes from minute 0 to minute 0 + 60 minutes.
  Measurement of patient's vital signs: blood pressure with a portable monitor every 15 minutes from t0 to t0 + 60 min
Any other hemodynamic and respiratory adverse event | The time of initiation of the ketamine or esketamine infusion defines the minute 0 time point of the study. The intensity of the psychodysleptic effects will be assessed by patients every 5 minutes from minute 0 to minute 0 + 60 minutes.
  Measurement of patient's vital signs : heart rate with a portable monitor every 15 minutes from t0 to t0 + 60 min
Any other hemodynamic and respiratory adverse event | The time of initiation of the ketamine or esketamine infusion defines the minute 0 time point of the study. The intensity of the psychodysleptic effects will be assessed by patients every 5 minutes from minute 0 to minute 0 + 60 minutes.
  Measurement of patient's vital signs : pulsed oxygen saturation with a portable monitor every 15 minutes from t0 to t0 + 60 min

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes-maritimes, France